CLINICAL TRIAL: NCT02046291
Title: Safety of Romiplostim (Nplate®) in Patients Who Have Failed to Achieve Platelet Engraftment Following Umbilical Cord Blood Transplant
Brief Title: Safety of Romiplostim (Nplate®) Following UCBT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012LS089; MT2012-17R (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Hematologic Malignancies
Keywords: umbilical cord transplant; acute leukemia; UCBT; Hodgkin's Lymphoma; Lymphoid Leukemia; Multiple Myeloma; Myeloid and Monocytic Leukemia; Non-Hodgkin's Lymphoma; Hematopoietic malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Hodgkin Disease; Leukemia, Lymphoid; Multiple Myeloma; Leukemia, Monocytic, Acute; Lymphoma, Non-Hodgkin | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Romiplostim treatment (Experimental): Romiplostim at the assigned dose will be administered subcutaneously (SQ) once a week for 6 weeks (i.e. 6 doses) unless platelet count exceeds 100 x 10^9/L and at least 4 doses of therapy were given.After the initial dose, subsequent doses will be administered within a window of +/- 3 days.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim at the assigned dose will be administered subcutaneously (SQ) once a week for 6 weeks. The dose will be assigned at the time of subject registration. This is a dose escalation to determine the maximum tolerated dose. The doses include 4 mcg/kg/dose, 6 mcg/kg/dose, 8 mcg/kg/dose, and 10 mcg/kg/dose.
  Other Names: Nplate

SUMMARY:
This is a single institution, phase I dose escalation study of weekly romiplostim post umbilical cord blood transplantation in patients who fail to achieve platelet engraftment by day +30. Engraftment is defined as a platelet count ≥ 20 x 109/L on 3 consecutive measurements without transfusion for 7 days. Romiplostim is administered at the assigned dose as 6 weekly injections beginning by day +42 post transplant. Up to 4 dose levels (4, 6, 8, and 10 mcg/kg/dose) will be evaluated with the maximum tolerated dose (MTD) of romiplostim determined by using the Continual Reassessment Method (CRM). The goal of this CRM will be to identify 1 of the 4 dose levels which corresponds to the desired maximum toxicity rate of 20% or less.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone a single or double umbilical cord blood transplant (UCBT) except those with primary myelofibrosis.

  * Those with acute leukemia must be in remission at the time of transplant
* Must have achieved neutrophil engraftment (defined as an ANC >500 for three consecutive days) and be off daily G-CSF prior to starting romiplostim. Intermittent G-CSF is allowed.
* Failure to achieve platelet engraftment (defined as platelet count ≥20x10^9/L on 3 consecutive measurements without transfusion for 7 days) by day +28 post UCBT
* Between day +28 and day +42 status post myeloablative or nonmyeloablative UCBT (single or double cord blood transplant)
* Age ≥ 18 years
* Adequate organ function within 7 days of enrollment defined as:

  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: SGOT and SGPT < 5 x upper limit of institutional normal (ULN)
* Women of child bearing potential agree to use effective contraception during therapy and for 4 months after completion of therapy
* Voluntary written consent

Exclusion Criteria:

* Known pregnancy - Pregnancy Category C: there are no adequate and well-controlled studies of romiplostim in pregnancy
* Recurrence of AML or myelodysplastic syndrome on bone marrow evaluation done within 21 days of enrollment
* Presence of clinically significant bone marrow fibrosis on the bone marrow examination immediately prior to UCBT
* Patients requiring more than one platelet transfusion per day
* History of an allergy to romiplostim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of romiplostim | Day +28 blood transplant (UCBT)
  Measured by number of patients who have failed to achieve platelet engraftment by day +28 after a myeloablative or nonmyeloablative umbilical cord blood transplant (UCBT)

SECONDARY OUTCOMES:
Platelet recovery | Day +28
  Average speed of platelet recovery in patients who have failed to achieve platelet engraftment.
Thrombocytopenia | Day +28
  Incidence of clinically significant bleeding episodes and number of platelet transfusions.
Bone marrow fibrosis | Day 100 post transplant
  Incidence of bone marrow fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, MSc, FRCPC, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States